CLINICAL TRIAL: NCT04793334
Title: Underlying Mechanisms of Obesity-induced Obstructive Sleep Apnea
Acronym: Slim-OSA
Status: Enrolling by invitation | Type: Observational
Sponsor: Brandon Nokes (Other)
Responsible Party: Sponsor-Investigator, Brandon Nokes, Post-doctoral fellow, Division of Pulmonary, Critical Care, Sleep Medicine, and Physiology, University of California, San Diego
Organization: University of California, San Diego (Other)
Other Study IDs: UCSD HRPP 191948
Record Dates: First submitted 2021-03-05; First posted 2021-03-11 (Actual); Last update posted 2024-05-29 (Actual); Status verified 2024-05

CONDITIONS: Obstructive Sleep Apnea; Obesity
MeSH Terms: conditions — Sleep Apnea, Obstructive; Obesity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Routine phlebotomy for blood gas analysis and exploratory biomarker assessment
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Obese + OSA: Inclusion Criteria:
  * Men and women
  * Ages >= 18-65 years old
  * BMI 35 kg/m2-above
  * Scheduled for sleeve gastrectomy (bariatric surgery)
  * OSA identified by PSG
  Exclusion Criteria:
  * Any cardiovascular, pulmonary or renal disease other than well-controlled hypertension or asthma.
  * Pregnancy
  * Currently smoking
  * Any respiratory disorder other than OSA or well controlled asthma
  * contraindication to MRI
  Interventions: Procedure: sleeve gastectomy
- Obese without OSA: Inclusion Criteria:
  * Men and women
  * Ages >= 18-65 years old
  * BMI 35kg/m2 and above
  * Scheduled for sleeve gastrectomy (bariatric surgery)
  * No OSA identified by PSG
  Exclusion Criteria:
  * Any cardiovascular, pulmonary or renal disease other than well-controlled hypertension or asthma.
  * Pregnancy
  * Currently smoking
  * Any respiratory disorder other than OSA or well controlled asthma
  * contraindication to MRI
  Interventions: Procedure: sleeve gastectomy

INTERVENTIONS:
Procedure: sleeve gastectomy — routine sleeve gastrectomy

SUMMARY:
Obesity is a common risk factor for the development of obstructive sleep apnea. However, not all subjects with obesity develop obstructive sleep apnea. This study will attempt to determine the mechanistic drivers between obesity and obstructive sleep apnea.

DETAILED DESCRIPTION:
Obstructive sleep apnea (OSA) is a highly prevalent disease with major neurocognitive and cardiovascular sequelae. Obesity is a major risk factor for OSA, but the underlying mechanisms remain unclear. Given the rising prevalence of obesity and the lack of adequate therapies for some afflicted patients, further mechanistic work is clearly required. Bariatric surgery is being done increasingly with compelling outcome data emerging; however, clinical response to weight loss is highly variable. In some patients, OSA is not present at baseline, despite morbid obesity, in other patients, OSA resolves following bariatric surgery, while other patients have persistence of OSA despite weight loss, and still other patients can experience re-emergence of OSA in long term follow-up studies after bariatric surgery. OSA can occur due to several major pathophysiological factors including pharyngeal anatomy, pharyngeal dilator muscle dysfunction, unstable ventilatory control, end- expiratory lung volume and arousal threshold. As a result considerable complexity exists in the obesity/OSA relationship, suggesting the need for further research. First, the investigators will perform a baseline evaluation of pathophysiological traits among obese people prior to weight loss surgery. Because some people will have OSA and some will not, the investigators will define the potential mechanisms underlying OSA and potential protective mechanisms among obese people without OSA (pharyngeal critical closing pressure Pcrit primary outcome). Second, the investigators will re-evaluate these same individuals from the standpoint of sleep study and pathophysiological traits six months following bariatric surgery after a variable degree of weight loss. The investigators anticipate that some OSA patients will have resolution of OSA whereas others will have persistence of disease. For non-OSA patients undergoing weight loss, the investigators will have a positive control group which will allow the investigators to account for non-specific effects of weight loss. This aim will allow the investigators to test the hypothesis that pharyngeal mechanics is the predominant mechanism whereby weight loss leads to improvement in OSA. Third, the investigators will perform magnetic resonance imaging during wakefulness at functional residual capacity, total lung capacity and residual volume on participants at baseline and 6months following bariatric surgery. This aim will allow the investigators to perform structure/function assessments in our participants, to define the impact of weight loss on pharyngeal anatomy, and to quantify the lung volume dependence of the upper airway before and after weight loss. The acquired data will also be used for computational modeling including dynamic assessment of pharyngeal function during tidal breathing. As a result of the proposed research, the investigators are confident that the investigators will gain major insights into the as yet unanswered question "why does obesity (sometimes) cause sleep apnea". This research will have major therapeutic implications as it will allow the investigators to individualize therapy for afflicted patients.

ELIGIBILITY:
Inclusion Criteria:

* - Men and women
* Ages >= 18-65 years old
* BMI 35 kg/m2--and above
* Scheduled for sleeve gastrectomy (bariatric surgery)

Exclusion Criteria:

* Any cardiovascular, pulmonary or renal disease other than well-controlled hypertension or asthma.
* Pregnancy
* Currently smoking
* Any respiratory disorder other than OSA or well controlled asthma
* contraindication to MRI

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Noting the inclusion and exclusion criteria above, we aim to recruit 110 patients, anticipating 20% drop out and a final n of 90. Further, we aim for to recruit 60 participants with OSA and 30 participants without OSA.
Sampling Method: Non-Probability Sample
Enrollment: 110 (Estimated)
Dates: Start 2021-03-20 (Actual); Primary Completion 2025-05-31 (Estimated); Study Completion 2026-05-31 (Estimated)

PRIMARY OUTCOMES:
muscle traits contributing to OSA in obesity - change is being assessed over time | Time point 1: Within 1 month of bariatric surgery, Time point 2: 6 months following bariatric surgery
  1. To measure upper airway collapsibility as well as the other traits (e.g. muscle responsiveness) in both groups. The traits can be measured during sleep using our well-validated research method that mimics transient upper airway obstruction and importantly, assesses the individual's response to hypoventilation
changes in pcrit after bariatric surgery | Time point 1: Within 1 month of bariatric surgery, Time point 2: 6 months following bariatric surgery
  2. We will reassess obese people with and without OSA following major weight loss (bariatric surgery). This aim will allow us to test the hypothesis that patients who experience improvement in OSA will be those with the greatest improvement in upper airway mechanics (Pcrit). The obese people without OSA undergoing weight loss will be a positive control group, which will allow us to exclude non-specific effects of weight loss.
MRI upper airway changes following bariatric surgery - change is being assessed over time | Time point 1: Within 1 month of bariatric surgery, Time point 2: 6 months following bariatric surgery
  3. To determine the anatomic correlates of upper airway collapsibility in both groups using magnetic resonance imaging during natural sleep.

SECONDARY OUTCOMES:
exploratory outcomes | Time point 1: Within 1 month of bariatric surgery, Time point 2: 6 months following bariatric surgery
  phlebotomy for ABG and transcriptomic assessments - change is being assessed over time

CONTACTS AND LOCATIONS:
Locations (1):
- UCSD - Altman Clinical Research Institute (ACTRI), La Jolla, California, United States